CLINICAL TRIAL: NCT02691390
Title: Exploration of the Potential Role of Anterior Cingulate (ACC) dTMS in Relapse to Alcohol Use
Brief Title: Deep Repetitive Transcranial Magnetic Stimulation for Alcohol Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Hadar Shalev, head of neuropsychiatric clinic soroka medical center, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sor040415ctil
Record Dates: First submitted 2016-02-07; First posted 2016-02-25 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (Experimental): alcoholics - dTMS group
  Interventions: Device: Active dTMS
- control group (Sham Comparator): alcoholics - sham group
  Interventions: Device: Sham dTMS

INTERVENTIONS:
Device: Active dTMS — dTMS to ACC
  Arms: study group
Device: Sham dTMS — SHAM - no stimulation
  Arms: control group

SUMMARY:
dTMS intervention to reduce recurrent alcohol abuse among alcohol users who are abstinent for at least 5 days.

DETAILED DESCRIPTION:
Phase 1: (up to 2 weeks), participants undergo a set of baseline assessments, including questionnaires, rating scales, and resting state functional magnetic resonance imaging (rsfMRI).

Phase 2, patients receive one of two treatments: High-frequency (10Hz, 100 trains of 3 sec with 15 sec inter train interval) dTMS targeting the ACC or sham stimulation for 30 min. Each treatment is preceded by provocation (pouring, holding and smelling the subject's favorite alcoholic beverage) designed to activate the relevant brain circuitry (provocation of symptoms may increase response rate to Deep TMS as was evident in the treatment of PTSD, cigarette smoking and OCD). dTMS sessions are conducted five times per week for 3 weeks, for a total of 15 sessions. A second scan that include rsfMRI and a risk-related decision-making task is conducted at the end of this phase.

Phase 3 includes 12 weeks of patients' follow-up, including clinical visits at weeks 1, 2, 4, 8 and 12 post treatment. During this phase, subjective and objective measures of alcohol use (self-report and analysis of urine samples for levels of ethyl glucuronide (EtG) and ethyl sulfate (EtS), respectively) are collected. Following completion of the main part by the individual, an "open label" treatment using the same parameters of the experiment is offer (regardless of treatment group).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65
* Current diagnosis of alcohol dependence
* Alcohol use in the past month
* Right handed (self-report)
* If female, negative urine pregnancy test
* If female, must either agree to practice an effective birth control method; agree to abstinence from intercourse; be surgically sterile or postmenopausal for at least one year

Exclusion Criteria:

* Currently pregnant or breastfeeding
* More than mild cognitive impairment, as determined by a score on the Montreal cognitive assessment (MoCA) <25.
* Current diagnosis of schizophrenia, bipolar disorder, or other psychotic disorder
* Use in the past 2 weeks of medication or illicit drug with known high pro-convulsant action, as self-reported, or detected using urine toxicology screening; and with accordance to the Physician best Judgment.
* Any history of clinically significant neurological disorders, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes (self-reported history).
* Any history of seizures other than febrile childhood seizures (self-reported history)
* Clinically significant hearing impairment
* Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces). Eligibility will be determined by the "MRI Safety Screening Questionnaire" and verified, if necessary, by a radiology consultant. Some of the patients that will be excluded from the imaging part of the study will be included in the clinical part.
* Any psychiatric, medical or social condition whether or not listed above, due to which, in the judgment of the investigators and after any consults if indicated, participation in the study is not in the best interest of the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Alcohol usage | 12 weeks post treatment
  The percentage of heavy drinking days (pHDD; 4+ alcohol units per women and 5+ for men, within one day) between the active and sham groups over the follow up period.

SECONDARY OUTCOMES:
Alcohol craving | 12 weeks post treatment
  The scores of the Penn alcohol craving scale (PACS) between the active and sham groups over the follow up period. The PACS is a 5-item questionnaire that measures the individual's alcohol craving in the past week, with each item scored on a scale between 0 and 6 (i.e., minimum value of 0 and maximum value of 30) and higher scores denote higher levels of craving.

OTHER OUTCOMES:
Modifications to brain volume | 3 weeks of treatment
  Changes to volumes (cm3) of brain areas that are implicated in alcohol abuse pathophysiology, as measured by MRI from pre- to post-treatment between the active and sham groups.
Modifications to functional connectivity | 3 weeks of treatment
  Changes to functional connectivity (correlation coefficient) of networks that are implicated in alcohol abuse pathophysiology, as measured by resting state fMRI from pre- to post-treatment between the active and sham groups
Modifications to blood-oxygen-level-dependent (BOLD) signal | 3 weeks of treatment
  Changes to blood-oxygen-level-dependent (BOLD) signal (arbitrary units) of brain areas that are implicated in alcohol abuse pathophysiology during behavioral tasks, as measured by fMRI following treatment between the active and sham groups.

IPD SHARING:
Plan to Share IPD: No